CLINICAL TRIAL: NCT01724372
Title: The Role of Antidepressants or Antipsychotics in Preventing Psychosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: The Zucker Hillside Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-094
Record Dates: First submitted 2012-11-01; First posted 2012-11-09 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2012-11

CONDITIONS: Psychotic Disorder
MeSH Terms: conditions — Psychotic Disorders | interventions — Antidepressive Agents; Fluoxetine; Antipsychotic Agents; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antidepressant (Experimental): Fluoxetine
  Interventions: Drug: Antidepressant
- Antipsychotic (Active Comparator): Aripiprazole
  Interventions: Drug: Antipsychotic

INTERVENTIONS:
Drug: Antidepressant
  Other Names: Fluoxetine
  Arms: Antidepressant
Drug: Antipsychotic
  Other Names: Aripiprazole
  Arms: Antipsychotic

SUMMARY:
This is a randomized, controlled pilot study comparing the antidepressant fluoxetine with the second generation antipsychotic aripiprazole in approximately 10 subjects aged 12-25 at risk for developing psychosis.

Our primary hypotheses are that compared to aripiprazole, fluoxetine will be better tolerated and will lead to greater improvement in symptoms at the end of 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 12-25 years of age (inclusive)
* Able to understand and speak English
* Have at least one sub-threshold positive psychotic symptom that is moderate, moderately severe, or severe

Exclusion Criteria:

* Lifetime diagnosis of an Axis I psychotic disorder: schizophreniform disorder; schizophrenia; schizoaffective disorder; bipolar disorder; or major depression with psychotic features
* Current psychosis
* Current diagnosis of Major Depressive Disorder, single episode or recurrent, severe without psychotic features
* Lifetime diagnosis of substance abuse or dependence (excluding nicotine)
* Current stimulant treatment
* Any significant medical condition that contra-indicates treatment with either aripiprazole or fluoxetine, including history of neurological, neuroendocrine or other medical condition known to affect the brain
* Estimated intelligence quotient < 70

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Attenuated positive, negative and general psychiatric symptoms | 6 months
  To compare fluoxetine and aripiprazole on the likelihood of and time to symptomatic improvement.

SECONDARY OUTCOMES:
Social and role functioning | 6 months
  To compare the effect of fluoxetine and aripiprazole on social and role functioning and subjective well-being in individuals at risk for schizophrenia.
Time to all-cause discontinuation. | 6 months
  To compare aripiprazole and fluoxetine on time to all-cause discontinuation or need to add another psychiatric medication.
Adverse effects | 6 months
  To compare aripiprazole and fluoxetine on the presence of associated rates of adverse effects.